CLINICAL TRIAL: NCT06874218
Title: Digital Analysis of Primary Teeth Crown Dimensions and Clinical Evaluation in a Sample of Egyptian Children
Acronym: Digital Analys
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Reham Abdelwahed Melegy, assistant lecture, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Digital Analysis of teeth; PED1-252299 (Registry Identifier: Research Ethics Committee Faculty of Dentistry)
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Primary Teeth Crown Dimensions in a Sample of Egyptian Children
Keywords: Teeth Dimensions; Digital Analysis; Egyptian Children

STUDY DESIGN:
Intervention Model Description: Digitally determine crown dimensions of primary teeth in a sample of Egyptian children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Primary Teeth Crown Dimensions in a Sample of Egyptian Children (Other): Digitally determine crown dimensions of primary teeth in a sample of Egyptian children
  Interventions: Device: prefabricated CAD-CAM Zirconia crowns according to Egyptian sizes.

INTERVENTIONS:
Device: prefabricated CAD-CAM Zirconia crowns according to Egyptian sizes. — compare prefabricated zirconia crowns according to the Egyptian crown sizes with the international standard zirconia crowns sizes for primary upper central incisors

SUMMARY:
The aim of this study will be conducted to:

1. Digitally determine crown dimensions of primary teeth in a sample of Egyptian children.
2. Clinical evaluation of prefabricated zirconia crowns according to the Egyptian sizes compared with the international standard zirconia crowns sizes for primary upper central incisors

DETAILED DESCRIPTION:
Currently, there is limited availability of primary tooth crown measurement for Egyptian children. SO, this study aims to digitally determine tooth crown dimensions of primary teeth in a group of Egyptian children and compare prefabricated zirconia crowns according to the Egyptian crown sizes with the international standard zirconia crowns sizes for primary upper central incisors.

ELIGIBILITY:
Inclusion Criteria:

* Children having normal fully erupted primary teeth and with no morphological variations.
* Children with no history of orthodontic or prosthodontic treatment.
* Children with normal overjet and overbite.
* Sound interproximal & buccal / lingual walls with or without minimal occlusal pits & fissure incipient caries.
* No previous interproximal & buccal / lingual restorations.
* Intact mesial and distal marginal ridge.

Exclusion Criteria:

* Children with gross carious lesions.
* Children with hypo-mineralization, hypoplasia and fracture primary teeth.
* Children with medical disabilities

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
crown dimensions of primary teeth in a sample of Egyptian children. | intra operative
  Digitally determine crown dimensions of primary teeth in a sample of Egyptian children using intraoral scanner and Digital measurements of teeth dimensions by Meshmixer analyzing software.

SECONDARY OUTCOMES:
Clinical evaluation of prefabricated zirconia crowns according to the Egyptian sizes compared with the international standard zirconia crowns sizes for primary upper central incisors. | intra operative
  Clinical evaluation of prefabricated zirconia crowns according to the Egyptian sizes compared with the international standard zirconia crowns sizes for primary upper central incisors by Modified United States Public Health Service (USPHS) criteria, and the gingival state near the primary performed crown will be assessed by using the Silness& Loe indices (1964) to record plaque index and gingival index.

CONTACTS AND LOCATIONS:
Overall Officials: Reham Abdelwahed Melegy, MSC, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
for patient privacy